CLINICAL TRIAL: NCT00193050
Title: Phase II Trial of Induction Chemotherapy With Weekly Gemcitabine, Epirubicin, Docetaxel as Primary Treatment of Locally Advanced or Inflammatory Breast Cancer Patients
Brief Title: Weekly Gemcitabine, Epirubicin, and Docetaxel in Locally Advanced or Inflammatory Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pharmacia and Upjohn (Industry); Eli Lilly and Company (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 51
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-09-21 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Epirubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): In the neoadjuvant setting, patients were administered gemcitabine (800 mg/m2 IV days 1 and 8), epirubicin (75 mg/m2 IV day 1), and docetaxel (30 mg/m2 IV days 1 and 8)repeated every 21 days for 4 cycles
  Patients then had either mastectomy or breast conservation surgery and pathologic treatment responses were assessed.
  After surgery, 4 cycles of adjuvant gemcitabine (1000 mg/m2 IV days 1 and 8) and docetaxel (35 mg/m2 IV days 1 and 8) were administered at 21 day intervals.
  After completion of chemotherapy, local regional radiation therapy and/or anti-estrogen therapy was administered per standard guidelines.
  Interventions: Drug: Gemcitabine; Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine
  Other Names: Gemzar
Drug: Epirubicin — Epirubicin
  Other Names: Ellence
Drug: Docetaxel — Docetaxel
  Other Names: Taxotere

SUMMARY:
Treatment strategies that include induction chemotherapy have several potential advantages: early initiation of systemic chemotherapy, in vivo assessment of response, and down-staging of both the primary tumor and regional lymphatic metastases, making breast conservation an option for many. The aim of the present study is to determine the efficacy and toxicity of induction combination chemotherapy with the triplet, gemcitabine, epirubicin, and docetaxel, in patients with locally advanced or inflammatory breast cancer. Clearly, it is in the upfront treatment as well as in the adjuvant treatment of breast cancer, that effective new agents and combination of agents are likely to have the greatest potential impact.

DETAILED DESCRIPTION:
Upon determination of eligibility, all patients will be receive:

Gemcitabine + Epirubicin + Docetaxel

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Adenocarcinoma of the breast confirmed by biopsy
* Female Patients >18 years of age
* Normal cardiac function
* Ability to perform activities of daily living with minimal assistance
* Chemotherapy naïve or have received prior chemotherapy > 5 years ago
* Adequate bone marrow, liver and kidney function
* Be informed of the investigational nature of this study
* Sign an informed consent form
* Sentinel lymph node and/or axillary dissection prior to enrollment

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Life expectancy of < than 6 months
* History of significant heart disease
* Prior chemotherapy or hormonal therapy
* Concurrent Trastuzumab therapy
* History of significant psychiatric disorders
* History of active uncontrolled infection

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2001-11; Primary Completion 2008-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A. Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Yardley DA, Peacock NW, Dickson NR, White MB, Vazquez ER, Foust JT, Grapski R, Hendricks LK, Scott WL, Hainsworth JD. A phase II trial of neoadjuvant gemcitabine, epirubicin, and docetaxel as primary treatment of patients with locally advanced or inflammatory breast cancer. Clin Breast Cancer. 2010 Jun;10(3):217-23. doi: 10.3816/CBC.2010.n.029. PMID 20497920
- See also: Published article in Clinical Breast Cancer — http://cigjournals.metapress.com/content/u57304468001h722/

RESULTS

PARTICIPANT FLOW:
Period: Neoadjuvant Treatment
Arm/Group | Intervention
Started | 110
Completed | 101
Not Completed | 9
Not completed — Lack of Efficacy | 2
Not completed — Intercurrent Illness | 3
Not completed — Physician Decision | 2
Not completed — Adverse Event | 2
Period: Surgery
Arm/Group | Intervention
Started | 103 (2 patients had surgery after 2 cycles of neoadjuvant treatment)
Completed | 103
Not Completed | 0
Period: Adjuvant
Arm/Group | Intervention
Started | 87 (16 patients never initiated postoperative adjuvant therapy)
Completed | 77
Not Completed | 10
Not completed — Physician Decision | 5
Not completed — Intercurrent Hospitalization | 3
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 110
Age, Continuous [Median (Full Range); unit: years] | 51 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 110

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response (pCR)
Description: For the purpose of this study, a Pathologic complete response (pCR) was defined as no evidence of residual invasive tumor in the breast (pT0). Residual ductal or lobular carcinoma in situ was not considered in pCR assessments. Percentage of participants who experienced pCR is reported.
Time Frame: 18 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 110
percentage of participants | 18 [11 to 26]

2. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to Treatment Failure (TTF) is defined as the minimum of the time from first date of treatment to the either of the following dates:
  * disease progression date (RECIST or clinical)
  * death date
  * treatment discontinuation
Time Frame: 69 months
Measure: Median (Full Range); unit: months
Groups:
- Intervention: In the neoadjuvant setting, patients were administered gemcitabine (800 mg/m2 IV days 1 and 8), epirubicin (75 mg/m2 IV day 1), and docetaxel (30 mg/m2 IV days 1 and 8)repeated every 21 days for 4 cycles
  Patients then had either mastectomy or breast conservation surgery and pathologic treatment responses were assessed.
  After surgery, 4 cycles of adjuvant gemcitabine (1000 mg/m2 IV days 1 and 8) and docetaxel (35 mg/m2 IV days 1 and 8) were administered at 21 day intervals.
  After completion of chemotherapy, local regional radiation therapy and/or anti-estrogen therapy was administered per standard guidelines.
  Gemcitabine: Gemcitabine
  Epirubicin: Epirubicin
  Docetaxel: Docetaxel
Arm/Group | Intervention
Number analyzed (Participants) | 110
months | 13 [1 to 53]

3. Secondary Outcome: Overall Survival (OS)
Description: Number of participants that are alive at 48th months
Time Frame: 48 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 110
Participants | 72

ADVERSE EVENTS:
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 38/110
Serious Adverse Events (participants affected / at risk) | 17/110
Other Adverse Events (participants affected / at risk) | 71/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=110)
Febrile Neutropenia (Infections and infestations) | 11 (15)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Anemia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1) — Fatal Legionnaire's disease
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=110)
Neutrophils (Blood and lymphatic system disorders) | 45 — Neutropenia
Platelets (Blood and lymphatic system disorders) | 19 — Thrombocytopenia
Hemoglobin (Blood and lymphatic system disorders) | 13 — Anemia
Nausea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 10
Diarrhea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.